CLINICAL TRIAL: NCT06646289
Title: An Open-label, Multicenter, Phase 2 Follow-on Study for Second Eye Treatment of Patients Previously Treated With a Recombinant Adeno-associated Virus Vector (AAV5 hRKp.RPGR) for Gene Therapy of Adults and Children With X-linked Retinitis Pigmentosa Owing to Defects in Retinitis Pigmentosa GTPase Regulator (RPGR)
Brief Title: A Follow-on Study for Second-Eye Treatment for Participants Previously Treated With Gene Therapy for X-Linked Retinitis Pigmentosa (XLRP)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 74765340RPG2001; 74765340RPG2001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2024-10-16; First posted 2024-10-17 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: X-Linked Retinitis Pigmentosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Participants will receive a dose of AAV5 hRKp.RPGR under the retina (low-dose or intermediate-dose) on Day 1 depending on the dosage administered in study MGT009 (NCT03252847) in the past. After receiving the treatment, participants will be assessed for safety.
  Interventions: Biological: AAV5-hRKp.RPGR
- Cohort 2 (Experimental): Participants will receive the treatment dose of AAV5 hRKp.RPGR under the retina (low-dose or intermediate-dose) on Day 1 in the second eye once the safety will be determined in Cohort 1.
  Interventions: Biological: AAV5-hRKp.RPGR
- Cohort 3 (Other): The participants who are not willing to undergo surgery or are not eligible for surgery will be assessed in this cohort. They will be assessed yearly until 5 years after their initial eye surgery in previous study MGT009.
  Interventions: Other: No intervention (Follow-Up assessment)

INTERVENTIONS:
Biological: AAV5-hRKp.RPGR — AAV5-hRKp.RPGR will be administered sub-retinally.
  Other Names: JNJ-74765340, botaretigene sparoparvovec
  Arms: Cohort 1; Cohort 2
Other: No intervention (Follow-Up assessment) — Participants will not receive any intervention and will undergo follow-up assessment.
  Arms: Cohort 3

SUMMARY:
The purpose of this study is to assess the safety and tolerability of subretinal delivery of Adeno-associated Virus Vector (AAV5 hRKp.RPGR) gene therapy in adults and children with X-linked retinitis pigmentosa.

ELIGIBILITY:
Inclusion Criteria:

* Have been treated with AAV5-hRKp.RPGR in study MGT009 and have completed or is currently enrolled in Study MGT010
* Must sign an informed consent form indicating that they understand the purpose and procedures of the study and is willing to participate in the study
* Willing to adhere to the protocol and long-term follow-up

Exclusion Criteria:

- There are no specific exclusion criteria to enroll in this study

Min Age: 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2030-10-24 (Estimated); Study Completion 2030-10-24 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AE) | From baseline up to 5.5 years
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the intervention. An AE can be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non investigational) product, whether or not related to that medicinal (investigational or non investigational) product.
Change from Baseline in Best Corrected Visual Acuity (BCVA) by Early Treatment Diabetic Retinopathy Study (ETDRS) Chart Letter Scores | Baseline, Months 12, 24, 36, 48 and 60
  Change from baseline in BCVA by ETDRS chart letter scores in monocular assessment of the second treated eye will be assessed. BCVA was measured using the ETDRS Scale (ranging from 0 to 100 letters) in the study eye. An increase in the number of letters read correctly means that vision has improved and vice-versa.
Change from Baseline in Low Luminance Visual Acuity (LLVA) by ETDRS Chart Letter Score | Baseline, Months 12, 24, 36, 48 and 60
  Change in LLVA by ETDRS chart letter scores from baseline in monocular assessment of second treated eye will be assessed. Visual function assessments included LLVA assessment in each eye by ETDRS letters. The letter score ranges from 0 (worse score) to 100 (best score), and a gain in LLVA from baseline indicates an improvement in visual acuity.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (3):
- United States (2):
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - University of Michigan Kellogg Eye Center, Ann Arbor, Michigan
- Moorfields Eye Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency